CLINICAL TRIAL: NCT04221711
Title: Safety and Efficacy of Repetitive Peripheral Magnetic Stimulation in Patients With Achilles Tendinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gesundheitszentrum Woergl (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RPS001
Record Dates: First submitted 2020-01-02; First posted 2020-01-09 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Achilles Tendinopathy
Keywords: Tendinopathy; Achilles; Repetitive Magnetic Stimulation
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Intervention Model Description: The study design was chosen to be a randomized, controlled trial.
Masking Description: Since blinding is not possible for patients, only the statistician will be blinded with respect to the treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Repetitive pulsed magnetic stimulation (Experimental): Patients randomized in this group will receive rPMS (80 milliTesla ; 2 Hertz; OMNITRON® promed; Healthfactories Holding GmbH) three times a week for a total of 12 weeks. Thereby they will be lying in a prone position or sitting for 20 minutes with the magnet coil positioned over the mid-portion of the affected Achilles tendon (manufactures instruction).
  Interventions: Device: Repetitive pulsed magnetic stimulation
- Eccentric Calf Muscle Training for Achilles Tendinopathy (Active Comparator): Two types of eccentric exercises will be used. The calf muscle will be eccentrically loaded both with the knee straight and with the knee bent. Each of the two exercises will include an increasing number of repetitions (1. Week, 2-3 weeks, 4-12 weeks) done in 3 sets (e.g. 3x15, 3x20, 3x30 repetitions). The patients will be informed that muscle soreness during the first 1 to 2 weeks of training was to be expected. Patients will receive a visual exercise protocol.
  Interventions: Procedure: Eccentric Calf Muscle Training for Achilles Tendinopathy

INTERVENTIONS:
Device: Repetitive pulsed magnetic stimulation — OMNITRON ProMed is a rPMS (repetitive peripheral magnetic stimulation) device used for deep stimulation of muscles and/or neurones (outside the brain). The energy is delivered by way of a special round treatment coil, whose cover material is tested for biocompatibility.
  The OMNITRON ProMed device produces a high-energy impulse field and stimulates tissue, in particular soft tissue, muscles and neurons, by means of repetitive peripheral magnetic stimulation (rPMS). Short, extremely strong magnetic fields in the microsecond range are emitted non-invasively. OMNITRON ProMed works with short-term energy emission at a peak power of up to 60 million watts and a magnetic field strength of up to 100 milliTesla.
  The intensity of treatment can be set between 20 and 100 %. The device automatically adjusts the magnetic field strength and the frequency of the pulses emitted depending on the intensity selected.
  For comfortable transport and application the product is compact and portable.
  Arms: Repetitive pulsed magnetic stimulation
Procedure: Eccentric Calf Muscle Training for Achilles Tendinopathy — Patients will be asked to stand with their full body weight on the injured leg. From an upright body position and standing with all body weight on the forefoot and the ankle joint in plantar flexion, the calf muscle is then loaded by having the patient slowly lower the heel beneath the forefoot. The calf muscle will only be loaded eccentrically, not concentric. Instead, the non-injured leg is used to get back to the start position. The first set of this exercise is performed in an upright position, followed by a second set with the knee bent to 45°. This regimen is performed 2x per day.
  The patients are told to go ahead with the exercise even if they experienced pain. However, they are told to stop if the pain becomes disabling.
  Arms: Eccentric Calf Muscle Training for Achilles Tendinopathy

SUMMARY:
With this prospective, randomized, controlled trial the investigators want to investigate effects of a prolonged repetitive Peripheral Magnetic Stimulation (rPMS) intervention on Achilles tendinopathy and compare it to a well established intervention. This may provide clinicians with a new, non-pharmacological, non-invasive, near painless approach to treat tendinopathy.

Although promising results with comparable devices exist, a direct and valid conclusion on the overall clinical performance of the investigational device cannot be drawn. This is mainly due to different treatment protocols used in the literature and due to the lack of insight in the technical documentation of comparable devices. Further, the applied magnetic fields vary in their amplitude, frequency, waveform and/or stimulation durations.

Therefore, the main goal of this clinical investigation is the collection of clinical data on the clinical performance of the investigational device. This clinical data will subsequently serve as a main source for the clinical evaluation of the medical device.

DETAILED DESCRIPTION:
Tendons are collagenous tissues that link muscle to bone, and in best case, a painless transmission of force allows voluntary movement over a life time. Although tendons show long time underestimated repair and remodelling capacities, some of them (e.g. the human patellar or Achilles tendon) remain quite prone to injury. To make things worse, tendinous tissue reveals incomplete healing capacities and treatments seem to be ineffective to avoid the high injury recurrence rate and/or the occurrence of chronic tendon pain. Thus, both elite and recreational athletes, as well as the non-sporting population or workplace employees often suffer from symptoms like tendon swelling, localized tenderness, activity related pain and impaired performance, also known as tendinopathy. Such pain-induced restriction of mobility frequently means the end of a sporting carrier, deteriorates the quality of life and patients have to live with all harmful consequences of physical inactivity. One tendon most commonly afflicted by this debilitating musculoskeletal injury is the Achilles tendon. Although it is the strongest tendon in our body, the prevalence for tendinopathy can be as high as 56% among certain athletes.

The repetitive peripheral magnetic stimulation (rPMS) works through a deep operating, focused and painless stimulation mechanism generated by pulsed magnetic fields. This intervention is already successfully in use to accelerate the healing of bone fractures and to enhance the healing of operated rotator cuff tears. Additionally, data on in vitro tendon cells indicate the positive effect of rPMS on tendon tissue by stimulating cell proliferation, up-regulating tendon-specific gene expression and releasing anti-inflammatory cytokines and growth factors. More interestingly, intervention studies on the healing of rotator cuff tendon-to-bone injuries in rat models show increases in tendon stiffness and modulus and enhanced collagen organization, and type I collagen expression after prolonged rPMS without showing adverse effects in any mechanical or histological property. These results strongly support the hypothesis that rPMS might be effective in treating Achilles tendinopathy in humans. This intervention might reduce pain and functional limitations, reverse tendon degenerative changes and increase the impaired tendon mechanical and material properties.

ELIGIBILITY:
Inclusion Criteria:

* Men and non-pregnant women aged 18-60 years
* Patients suffering from a gradually evolving painful condition in the Achilles tendon located at the midportion for at least 12 weeks (Diagnosis based on clinical examination showing a painful thickening of the Achilles tendon located at a level of 2 to 6cm above the tendon insertion, and confirmed by ultrasonography: local thickening of the tendon, irregular tendon structure with hypoechoic areas and irregular fiber orientation).
* VISA-A score less than 65 at baseline.
* Be informed of the nature of the study and provide written informed consent.

Exclusion Criteria:

* Clinical suspicion of insertional disorders (pain at the site of the insertion of the Achilles tendon on the calcaneum)
* Concomitant or previous participation in a clinical investigation within the last 3 months (wash out) prior to study inclusion
* Clinical suspicion of an Achilles tendon rupture.
* Suspicion of internal disorders: spondylarthropathy, gout, hyperlipidemia, Rheumatoid Arthritis and sarcoidosis.
* Severe foot deformity
* Condition that prevents the patients from executing an active exercise program
* Pregnant or lactating females
* History of treatment with corticosteroids, estrogens, long term quinolone antibiotics, and cholesterol drugs
* Persons with electronic implants (e.g. pacemaker, cochlear implants, drug pump, deep brain stimulator, etc.)
* Patients with organ transplants
* Patients with closed, circular metal implants (e.g. subdermal implants, etc.)
* Epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09-04 (Estimated); Primary Completion 2021-09-04 (Estimated); Study Completion 2021-09-04 (Estimated)

PRIMARY OUTCOMES:
Change of the experience of pain and functionality with the Victorian Institute of Sports Assessment questionnaire (VISA-A) | "Week 0", "Week 12"
  Change of the experience of pain and functionality as assessed by the Victorian Institute of Sports Assessment questionnaire (VISA-A). The VISA-A questionnaire is a validated questionnaire with good test-retest, intra-rater and inter-rater reliability and is especially designed for patients with Achilles tendinopathy. The maximum score that can be achieved on the question is 100, and would be the score of person who is completely asymptomatic. A lower score indicates more symptoms and greater limitation of physical activity.
Change of the experience of pain at exertion as assessed by the Visual Analogue Scale (VAS) | "Week 4", "Week 12"
  Psychometric response scale with continuous aspect (Visual Analogue Scale (VAS)). 0 means low ("no pain"), 100 means high (Pain as bad as could possibly be).
Percentage of participants with an anticipated adverse event of special interest | "Week 4"
  Percentage of participants with an anticipated adverse event of special interest (muscle twitching, local warming and initial pain excitement). The occurrence of the expected side-effects is not definitely clear based on literature and pre-clinical investigations.

SECONDARY OUTCOMES:
Change of the experience of pain and functionality with the Victorian Institute of Sports Assessment questionnaire (VISA-A) | "Week 0", "Week 2"
  Change of the experience of pain and functionality as assessed by the Victorian Institute of Sports Assessment questionnaire (VISA-A). The VISA-A questionnaire is a validated questionnaire with good test-retest, intra-rater and inter-rater reliability and is especially designed for patients with Achilles tendinopathy. The maximum score that can be achieved on the question is 100, and would be the score of person who is completely asymptomatic. A lower score indicates more symptoms and greater limitation of physical activity.
Change of the experience of pain and functionality with the Victorian Institute of Sports Assessment questionnaire (VISA-A) | "Week 0", "Week 4"
  Change of the experience of pain and functionality as assessed by the Victorian Institute of Sports Assessment questionnaire (VISA-A). The VISA-A questionnaire is a validated questionnaire with good test-retest, intra-rater and inter-rater reliability and is especially designed for patients with Achilles tendinopathy. The maximum score that can be achieved on the question is 100, and would be the score of person who is completely asymptomatic. A lower score indicates more symptoms and greater limitation of physical activity.
Change of the experience of pain and functionality with the Victorian Institute of Sports Assessment questionnaire (VISA-A) | "Week 0", "Week 6"
  Change of the experience of pain and functionality as assessed by the Victorian Institute of Sports Assessment questionnaire (VISA-A). The VISA-A questionnaire is a validated questionnaire with good test-retest, intra-rater and inter-rater reliability and is especially designed for patients with Achilles tendinopathy. The maximum score that can be achieved on the question is 100, and would be the score of person who is completely asymptomatic. A lower score indicates more symptoms and greater limitation of physical activity.
Change of the experience of pain and functionality with the Victorian Institute of Sports Assessment questionnaire (VISA-A) | "Week 0", "Week 8"
  Change of the experience of pain and functionality as assessed by the Victorian Institute of Sports Assessment questionnaire (VISA-A). The VISA-A questionnaire is a validated questionnaire with good test-retest, intra-rater and inter-rater reliability and is especially designed for patients with Achilles tendinopathy. The maximum score that can be achieved on the question is 100, and would be the score of person who is completely asymptomatic. A lower score indicates more symptoms and greater limitation of physical activity.
Change of the experience of pain and functionality with the Victorian Institute of Sports Assessment questionnaire (VISA-A) | "Week 0", "Week 24"
  Change of the experience of pain and functionality as assessed by the Victorian Institute of Sports Assessment questionnaire (VISA-A). The VISA-A questionnaire is a validated questionnaire with good test-retest, intra-rater and inter-rater reliability and is especially designed for patients with Achilles tendinopathy. The maximum score that can be achieved on the question is 100, and would be the score of person who is completely asymptomatic. A lower score indicates more symptoms and greater limitation of physical activity.
Change of the experience of pain at exertion with Visual Analogue Scale (VAS) | "Week 0", "Week 2"
  Psychometric response scale with continuous aspect (Visual Analogue Scale (VAS)). 0 means low ("no pain"), 100 means high (Pain as bad as could possibly be).
Change of the experience of pain at exertion with Visual Analogue Scale (VAS) | "Week 0", "Week 4"
  Psychometric response scale with continuous aspect (Visual Analogue Scale (VAS)). 0 means low ("no pain"), 100 means high (Pain as bad as could possibly be).
Change of the experience of pain at exertion with Visual Analogue Scale (VAS) | "Week 0", "Week 6"
  Psychometric response scale with continuous aspect (Visual Analogue Scale (VAS)). 0 means low ("no pain"), 100 means high (Pain as bad as could possibly be).
Change of the experience of pain at exertion with Visual Analogue Scale (VAS) | "Week 0", "Week 8"
  Psychometric response scale with continuous aspect (Visual Analogue Scale (VAS)). 0 means low ("no pain"), 100 means high (Pain as bad as could possibly be).
Change of the experience of pain at exertion with Visual Analogue Scale (VAS) | "Week 0", "Week 24"
  Psychometric response scale with continuous aspect (Visual Analogue Scale (VAS)). 0 means low ("no pain"), 100 means high (Pain as bad as could possibly be).
Patient Satisfaction: Psychometric response scale with Visual Analogue Scale (VAS). | "Week 0"
  Psychometric response scale with continuous aspect (Visual Analogue Scale (VAS)). 0 means low ("not satisfied at all"), 100 means high (Satisfaction could not be higher).
Patient Satisfaction: Psychometric response scale with Visual Analogue Scale (VAS). | "Week 2"
  Psychometric response scale with continuous aspect (Visual Analogue Scale (VAS)). 0 means low ("not satisfied at all"), 100 means high (Satisfaction could not be higher).
Patient Satisfaction: Psychometric response scale with Visual Analogue Scale (VAS). | "Week 4"
  Psychometric response scale with continuous aspect (Visual Analogue Scale (VAS)). 0 means low ("not satisfied at all"), 100 means high (Satisfaction could not be higher).
Patient Satisfaction: Psychometric response scale with Visual Analogue Scale (VAS). | "Week 6"
  Psychometric response scale with continuous aspect (Visual Analogue Scale (VAS)). 0 means low ("not satisfied at all"), 100 means high (Satisfaction could not be higher).
Patient Satisfaction: Psychometric response scale with Visual Analogue Scale (VAS). | "Week 8"
  Psychometric response scale with continuous aspect (Visual Analogue Scale (VAS)). 0 means low ("not satisfied at all"), 100 means high (Satisfaction could not be higher).
Patient Satisfaction: Psychometric response scale with Visual Analogue Scale (VAS). | "Week 12"
  Psychometric response scale with continuous aspect (Visual Analogue Scale (VAS)). 0 means low ("not satisfied at all"), 100 means high (Satisfaction could not be higher).
Patient Satisfaction: Psychometric response scale with Visual Analogue Scale (VAS). | "Week 24"
  Psychometric response scale with continuous aspect (Visual Analogue Scale (VAS)). 0 means low ("not satisfied at all"), 100 means high (Satisfaction could not be higher).
Change of Achilles transverse thickness | "Week 0", "Week 6"
  Maximum thickness will be recorded in the midportion of the affected Achilles tendon
Change of Achilles transverse thickness | "Week 0", "Week 12"
  Maximum thickness will be recorded in the midportion of the affected Achilles tendon
Change of Neovascularization in the Achilles tendon | "Week 0", "Week 4"
  Doppler activity measured with real time ultrasonography in a longitudinal and sagittal view.
Change of Neovascularization in the Achilles tendon | "Week 0", "Week 12"
  Doppler activity measured with real time ultrasonography in a longitudinal and sagittal view.
Usability, graded on a scale from 1 to 5 (1 means low usability, 5 means high usability) | "Week 2"
  The usability characteristics contribute to the summative evaluation of the usability of the device under investigation. 1 means low usability, 5 means high usability.
Usability, graded on a scale from 1 to 5 (1 means low usability, 5 means high usability) | "Week 8"
  The usability characteristics contribute to the summative evaluation of the usability of the device under investigation. 1 means low usability, 5 means high usability.
Usability, graded on a scale from 1 to 5 (1 means low usability, 5 means high usability) | "Week 12"
  The usability characteristics contribute to the summative evaluation of the usability of the device under investigation. 1 means low usability, 5 means high usability.
Percentage of participants with an anticipated adverse event of special interest. | "Week 0"
  The percentage of participants with an anticipated adverse event of special interest (muscle twitching, local warming and initial pain excitement). The occurrence of the expected side-effects is not definitely clear based on literature and pre-clinical investigations.
Percentage of participants with an anticipated adverse event of special interest. | "Week 2"
  The percentage of participants with an anticipated adverse event of special interest (muscle twitching, local warming and initial pain excitement). The occurrence of the expected side-effects is not definitely clear based on literature and pre-clinical investigations.
Percentage of participants with an anticipated adverse event of special interest. | "Week 6"
  The percentage of participants with an anticipated adverse event of special interest (muscle twitching, local warming and initial pain excitement). The occurrence of the expected side-effects is not definitely clear based on literature and pre-clinical investigations.
Percentage of participants with an anticipated adverse event of special interest. | "Week 8"
  The percentage of participants with an anticipated adverse event of special interest (muscle twitching, local warming and initial pain excitement). The occurrence of the expected side-effects is not definitely clear based on literature and pre-clinical investigations.
Percentage of participants with an anticipated adverse event of special interest. | "Week 12"
  The percentage of participants with an anticipated adverse event of special interest (muscle twitching, local warming and initial pain excitement). The occurrence of the expected side-effects is not definitely clear based on literature and pre-clinical investigations.
Percentage of participants with an anticipated adverse event of special interest. | "Week 24"
  The percentage of participants with an anticipated adverse event of special interest (muscle twitching, local warming and initial pain excitement). The occurrence of the expected side-effects is not definitely clear based on literature and pre-clinical investigations.

CONTACTS AND LOCATIONS:
Locations (1):
- Gesundheitszentrum Woergl, Wörgl, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No